CLINICAL TRIAL: NCT00973921
Title: Comparison of StentOptimizer - an Angiography-based Post Deployment Stent Analysis Application With IntraVenous Ultrasound and 2D Quantitative Coronary Angiography for Post Deployment Stent Analysis
Brief Title: Comparison of StentOptimizer With IntraVenous Ultrasound and 2D Quantitative Coronary Angiography
Status: Completed | Type: Observational
Sponsor: Paieon Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Paieon-Columbia-SO
Record Dates: First submitted 2009-09-06; First posted 2009-09-09 (Estimated); Results first posted 2014-04-11 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-03

CONDITIONS: Coronary Artery Disease
Keywords: Stent; under-expansion; StentOp; StentOptimizer; IVUS; IC-PRO; image enhancement
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stent deployment evaluation: The study group consisted of patients that underwent IVUS guided stent implantation. Stent deployment evaluation was done with the experimental StentOptimizer as well as IVUS and QCA.

SUMMARY:
The primary objective of this study is to determine the diagnostic efficiency and accuracy of using the StentOptimizer. The ability of StentOptimizer to influence post deployment treatment strategy will be assessed and compared to the IVUS system. In addition, the correlation of diameter measurements between the StentOptimizer, IVUS and 2D QCA will be assessed. The StentOptimizer software, IVUS and 2D QCA were all part of the clinical procedure outside the study. The analysis of post deployment treatment decisions and diameter measurements using those modalities retrospectively make this an observational study.

DETAILED DESCRIPTION:
Stent under-expansion is defined as the minimum stent area by itself or compared with a predefined reference. It plays a role in the pathogenesis of adverse events following stent deployment. Stent under-expansion has been a consistent finding in IVUS reports of acute or subacute BMS or DES thrombosis.

Post intervention imaging can determine whether there is adequate stent expansion. Currently the only available tool for evaluation of properness of stent deployment is intravascular ultrasound (IVUS). IVUS procedure is invasive, labor intensified, associated with radiation and contrast media use, and is not free of complications. In many medical centers, IVUS is not used routinely because of lack of knowledge and expertise in reading it, and it's relatively high price.

The StentOptimizer is an angiography based software tool aimed to enhance visualization of deployed stents and to provide the physician with quantitative data regarding stent dimensions. The StentOptimizer is part of an image acquisition and processing software system (IC-Pro), designed as an add-on to conventional X-ray angiography systems.

An enhanced stent image is produced using the radiopaque markers of the delivery balloon from several frames (minimum 20). The result is a still image of the stent with enhanced edges and the region of interest around it

ELIGIBILITY:
Inclusion Criteria:

1. Percutaneous coronary intervention indicated clinically.
2. IVUS used as part of the standard procedure.
3. Subject must be >=40 yrs.
4. Subject must provide written informed consent.

Exclusion Criteria:

1. Low image quality as determined by the investigator.
2. Subject is pregnant or nursing.
3. Acute ST segment elevation myocardial infarction (STEMI) that has not been stabilized.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients that underwent IVUS guided stent implantation in the institution.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giora Weisz, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Coronary Stenting Evaluation With IVUS: The study group consisted of patients who were scheduled for coronary artery stent placement procedures in which stent deployment evaluations with Intravascular Ultrasound (IVUS), Quantitative Coronary Angiography (QCA) and StentOptimizer (SO) software were clinically indicated.
Period: Overall Study
Arm/Group | Coronary Stenting Evaluation With IVUS
Started | 40
Completed | 31
Not Completed | 9
Not completed — IVUS results were not available | 9

BASELINE CHARACTERISTICS:
Arm/Group | Coronary Stenting Evaluation With IVUS
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: The Accuracy (Percent of Correct Decisions) of Post-dilatation Decisions Based on the Stent Optimizer (SO) Software, With IVUS as Gold Standard.
Description: IVUS was used as a gold standard to decide if a stent required post dilatation or not. Independently and blindly, The SO software was used to determine the same decisions. The accuracy of SO was determined as the percentage of correct decisions compared to the gold standard.
Time Frame: On the procedure day
Population: Total of 40 consecutive patients who underwent PCI with stent implantation were enrolled. Only 31 of them had analyzable IVUS results.
Measure: Number; unit: percentage of correct decisions by SO
Arm/Group | Coronary Stenting Evaluation With IVUS
Number analyzed (Participants) | 31
percentage of correct decisions by SO | 100
Statistical Analysis 1: Comparison: Coronary Stenting Evaluation With IVUS; The 95% confidence Interval (CI) of the primary outcome has been calculated using the Wilson method of estimating the CI of a single proportion; Test type: Superiority or Other; p < 0.01, Wilson; Proportion = 1.0, 95% CI 2-sided [0.86 to 1.0]

2. Secondary Outcome: Correlation of Stent Diameter Measurements Between the StentOptimizer and IVUS .
Description: The mean difference between stent diameter measurements at the narrowest point (Minimum Stent Diameter) by SO and by IVUS.
Time Frame: On day of procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Coronary Stenting Evaluation With IVUS
Number analyzed (Participants) | 31
mm | 0.1 (0.4)
Statistical Analysis 1: Comparison: Coronary Stenting Evaluation With IVUS; Test type: Superiority or Other; p < 0.0001, Bland Altman; Correlation coefficient = 0.74

3. Primary Outcome: The Accuracy (Percent of Correct Decisions) of Post-dilatation Decisions Based on QCA Analysis, With IVUS as Gold Standard.
Description: IVUS was used as a gold standard to decide if a stent required post dilatation or not. Independently and blindly, QCA analysis was used to determine the same decisions. The accuracy of SO was determined as the percentage of correct decisions compared to the gold standard.
Time Frame: On procedure day
Population: as for outcome 1
Measure: Number; unit: percentage of correct decision by QCA
Arm/Group | Coronary Stenting Evaluation With IVUS
Number analyzed (Participants) | 31
percentage of correct decision by QCA | 74.2

4. Secondary Outcome: Correlation of Stent Diameter Measurements Between the QCA and IVUS .
Description: The mean difference between stent diameter measurements at the narrowest point (Minimum Stent Diameter) by QCA and by IVUS
Time Frame: On day of procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Coronary Stenting Evaluation With IVUS
Number analyzed (Participants) | 31
mm | 0.3 (0.4)
Statistical Analysis 1: Comparison: Coronary Stenting Evaluation With IVUS; Test type: Superiority or Other; p = 0.0034, Bland-Altman; Correlation coefficient = 0.5

ADVERSE EVENTS:
Arm/Group | Coronary Stenting Evaluation With IVUS
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

LIMITATIONS AND CAVEATS:
This is a relatively small study designed to evaluate the procedural decision about post-deployment dilatation not powered to evaluate the outcome of patients. The operator decision of his post-dilatation strategy was qualitative.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No